CLINICAL TRIAL: NCT00000744
Title: A Randomized, Prospective, Double-Blind Study Comparing Fluconazole With Placebo for Primary and Secondary Prophylaxis of Mucosal Candidiasis in HIV-Infected Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Treatment
Other Study IDs: CPCRA 010; 11562 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Candidiasis; Candidiasis, Esophageal; HIV Infections
Keywords: Fluconazole; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Candidiasis
MeSH Terms: conditions — Candidiasis; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Fluconazole

INTERVENTIONS:
Drug: Fluconazole

SUMMARY:
To compare the efficacy of fluconazole versus placebo for the prevention of Candida esophagitis and vaginal/oropharyngeal candidiasis, including a comparison of the development of clinical resistance.

Fluconazole has been shown to be effective in preventing or suppressing candidiasis in HIV-negative women. An increasing likelihood of oral and esophageal candidiasis in conjunction with progressive immunosuppression raises the question of the potential role of prophylactic antifungal therapy in high-risk persons.

DETAILED DESCRIPTION:
Fluconazole has been shown to be effective in preventing or suppressing candidiasis in HIV-negative women. An increasing likelihood of oral and esophageal candidiasis in conjunction with progressive immunosuppression raises the question of the potential role of prophylactic antifungal therapy in high-risk persons.

Four hundred HIV-infected women are randomized to receive fluconazole or placebo weekly for up to 2 years. Patients undergo follow-up every 3 months or more often if signs and symptoms of mucosal candidiasis occur.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Evidence of HIV infection.
* CD4+ count <= 300 cells/mm3 or <= 20 percent of total lymphocyte count.
* Reasonably good health with a life expectancy of at least 6 months.
* Pelvic exam including Pap smear or colposcopy performed within the past 90 days.

Prior Medication:

Allowed:

* Topical or systemic treatment or prophylaxis with an antifungal agent.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Current diagnosis of Candida esophagitis.
* Known intolerance to azoles.

Concurrent Medication:

Excluded:

* Systemic treatment or prophylaxis with an antifungal agent.

Patients with the following prior conditions are excluded:

* Past history of Candida esophagitis.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Study Completion 1995-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P Schuman, Study Chair; L Capps, Study Chair
Locations (16):
- United States (16):
  - Community Consortium of San Francisco, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Wilmington Hosp / Med Ctr of Delaware, Wilmington, Delaware
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Addiction Research and Treatment Corp, Brooklyn, New York
  - Clinical Directors Network of Region II, New York, New York
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Schuman P, Capps L, Peng G, Vazquez J, el-Sadr W, Goldman AI, Alston B, Besch CL, Vaughn A, Thompson MA, Cobb MN, Kerkering T, Sobel JD. Weekly fluconazole for the prevention of mucosal candidiasis in women with HIV infection. A randomized, double-blind, placebo-controlled trial. Terry Beirn Community Programs for Clinical Research on AIDS. Ann Intern Med. 1997 May 1;126(9):689-96. doi: 10.7326/0003-4819-126-9-199705010-00003. PMID 9139554
- [Background] Capps L, Peng G, Doyle M, El-Sadr W, Neaton JD. Sexually transmitted infections in women infected with the human immunodeficiency virus. Terry Beirn Community Programs for Clinical Research on AIDS (CPCRA). Sex Transm Dis. 1998 Sep;25(8):443-7. doi: 10.1097/00007435-199809000-00012. PMID 9773440
- [Background] Vazquez JA, Sobel JD, Peng G, Steele-Moore L, Schuman P, Holloway W, Neaton JD. Evolution of vaginal Candida species recovered from human immunodeficiency virus-infected women receiving fluconazole prophylaxis: the emergence of Candida glabrata? Terry Beirn Community Programs for Clinical Research in AIDS (CPCRA). Clin Infect Dis. 1999 May;28(5):1025-31. doi: 10.1086/514746. PMID 10452629
- [Background] Vazquez JA, Peng G, Sobel JD, Steele-Moore L, Schuman P, Holloway W, Neaton JD. Evolution of antifungal susceptibility among Candida species isolates recovered from human immunodeficiency virus-infected women receiving fluconazole prophylaxis. Clin Infect Dis. 2001 Oct 1;33(7):1069-75. doi: 10.1086/322641. Epub 2001 Sep 5. PMID 11528582